CLINICAL TRIAL: NCT00280046
Title: Effect of Biphasic Insulin Aspart 30 on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Effect of Biphasic Insulin Aspart 30 on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1554
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart

SUMMARY:
This trial was conducted in Russian Federation. This trial aimed for a comparison of the effect on glycemic control in subjects with type 2 diabetes of three different treatment regimens: biphasic insulin aspart 30 thrice daily, biphasic insulin aspart 30 twice daily in combination with metformin and treatment with oral anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, currently treated with one or more oral hypoglycemic agent
* HbA1c: At least 8.0%

Exclusion Criteria:

* Impaired hepatic, renal or cardiac function

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2003-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 16 weeks of treatment

SECONDARY OUTCOMES:
Self-measured 7-point capillary plasma glucose profile
Change in body weight
Incidence of hypoglycaemic episodes and adverse events
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (11):
- Russia (11):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Belgorod
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Khabarovsk
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Omsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Vladivostok
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yekaterinburg

REFERENCES:
- [Result] Ushakova O, Sokolovskaya V, Morozova A, Valeeva F, Zanozina O, Sazonova O, Zhadanova E, Starceva M, Kazakova E, Saifullina M, Shapiro I, Tarasov A, Al-Tayar B, Starkova N. Comparison of biphasic insulin aspart 30 given three times daily or twice daily in combination with metformin versus oral antidiabetic drugs alone in patients with poorly controlled type 2 diabetes: a 16-week, randomized, open-label, parallel-group trial conducted in russia. Clin Ther. 2007 Nov;29(11):2374-84. doi: 10.1016/j.clinthera.2007.11.017. PMID 18158078
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com